CLINICAL TRIAL: NCT02410135
Title: Myrbetriq™ (Mirabegron) to Improve Disordered Sleep in Subjects With Lower Urinary Tract Symptoms (LUTS)
Status: Completed | Type: Observational
Sponsor: Southern Illinois University (Other)
Collaborators: Astellas Scientific & Medical Affairs, Inc. (Industry); Sisters of the Third Order of St. Francis (Other)
Responsible Party: Sponsor
Other Study IDs: MYRB-14B03
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2018-09

CONDITIONS: Lower Urinary Tract Symptoms; Nocturia
Keywords: Lower Urinary Tract Symptoms; Sleep Disturbance
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Nocturia; Parasomnias | interventions — mirabegron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with symptomatic LUTS and disordered sleep: Patients exhibiting symptoms of LUTS and disordered sleep and who meet all inclusion/exclusion criteria will be prescribed Mirabegron for 12 weeks.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — 25 mg PO per day for four weeks. if tolerated then uptitrated to 50 mg PO per day for the remaining 8 weeks
  Other Names: Myrbetriq

SUMMARY:
The objective of this exploratory pilot study is to assess whether Mirabegron (Myrbetriq™) will improve the quality of sleep and Lower Urinary Tract Symptoms (LUTS) in men and women presenting with LUTS and disordered sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Subject is willing and able to complete the micturition diary and sleep questionnaires correctly.
3. Symptoms of overactive bladder (OAB) (urinary frequency and urgency with or without urgency incontinence) for at least 3 months, with an IPSS ≥ 12.
4. Moderate sleep disturbance with a mean score on the Jenkins Scale > 7.
5. Micturitions/24 hrs ≥ 8; total excretory volume of <3L.
6. Washout period of 2 weeks for any drugs not listed in the exclusions.

Exclusion Criteria:

1. Subject is using prohibited medications which cannot be stopped safely at the screening visit. Subject is excluded if using restricted medications not meeting protocol-specified criteria:

   (i) Phytotherapy for benign prostatic hypertrophy (BPH) or a 5-alpha reductase inhibitor within 3 months.

   (ii) Alpha blocker within 2 weeks. (iii) Taken an oral alpha agonist, tricyclic antidepressants, and anticholinergic or cholinergic medication within 2 weeks of the first screening visit with the following exception: topical anticholinergic eye drops used for glaucoma or inhaled anti-cholinergic used for chronic obstructive pulmonary disease (COPD).

   (iv) Taken an estrogen, androgen, or any drug producing androgen suppression, or anabolic steroids within 3 months.
2. Post void residual volume > 350 mL.
3. Female subject is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential is sexually active and not practicing a highly reliable method of birth control.
4. Subject has neurogenic bladder.
5. Any prior invasive intervention for LUTS (including bladder paralytics such as botulin toxin)
6. Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the investigator (for female subjects confirmed by a cough provocation test).
7. Subject has an indwelling catheter or practices intermittent self-catheterization.
8. Known primary neurologic conditions such as multiple sclerosis, Parkinson's disease, diabetic neuropathy or any neurological diseases known to affect bladder function.
9. Subject has evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs.
10. Two documented independent urinary tract infections of any type in the past year.
11. Patient with a diagnosed sleep disorder (ie. Obstructive Sleep Apnea) undergoing evaluation and treatment requiring change in care within 30 days of screening visit.
12. Subject has moderate to severe hepatic impairment [ALT (SGPT), AST (SGOT) or GGT value greater than 3 times the upper limit of normal in the clinical center lab; confirmed on a second measurement].
13. Subject has severe renal impairment or End Stage Renal disease (i.e., creatinine greater than 2.0 mg/dl).
14. PSA (prostate specific antigen) level greater than 10 ng/ml at the first screening visit (if male).
15. Subject has severe uncontrolled hypertensionas defined by a systolic pressure ≥180 mmHg and/or diastolic pressure ≥120 mmHg.
16. Subject has a clinically significant abnormal ECG or has a known history of QT prolongation or currently taking medication known to prolong the QT interval.
17. Subject has a known or suspected hypersensitivity to Mirabegron or any of the inactive ingredients.
18. Subject has a concurrent malignancy or history of cancer (except noninvasive skin cancer) within the last 5 years prior to screening. Men with a history of prostate cancer regardless of curability are not eligible.
19. Subject has been treated with an experimental device within 30 days or received an experimental agent within the longer of 30 days or five half-lives.
20. Unable to follow protocol directions due to organic brain or psychiatric disease.
21. History of alcoholism or any other substance abuse, which, in the opinion of the investigator, would affect compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with lower urinary tract symptoms and sleep disturbance
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
• Improvement from baseline on the PROMIS Sleep Disturbance scale at the 12 week follow-up. | 12 weeks
• Improvement from baseline in the number micturitions/24 hours at the 12 week follow-up. | 12 weeks

SECONDARY OUTCOMES:
• Improvement from baseline on the Jenkins sleep scale at the 12 week follow-up. | 12 weeks
• Improvement of nocturia (nocturnal voiding) based on the amount of voids that disrupt patient sleep in the voiding diary. | 12 weeks

OTHER OUTCOMES:
• Improvement from baseline on the International Prostate Symptom Score (IPSS)/American Urological Society Symptom Index (AUA-SI) scale at the 12 week follow-up. | at 12 week follow-up
  exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Kevin McVary, MD, Principal Investigator — Southern Illinois University
Locations (1):
- SIUSOM - Division of Urology, Springfield, Illinois, United States